CLINICAL TRIAL: NCT01150630
Title: Randomized Phase II-III Trial of Peri- or Post-Operative Chemotherapy in Resectable Pancreatic Adenocarcinoma
Brief Title: Gemcitabine, Cisplatin, Epirubicin, and Capecitabine in Treating Patients With Stage I-II Resectable Pancreatic Cancer
Acronym: PACT-15
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Michele Reni, MD, IRCCS San Raffaele
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000675485; PACT-15 (Other: IRCCS San Raffaele); 2010-019942-23 (EudraCT Number)
Record Dates: First submitted 2010-06-24; First posted 2010-06-25 (Estimated); Last update posted 2017-09-01 (Actual); Status verified 2017-08

CONDITIONS: Pancreatic Cancer
Keywords: adenocarcinoma of the pancreas; stage I pancreatic cancer; stage II pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Capecitabine; Cisplatin; Epirubicin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- adjuvant PEXG (Experimental): cisplatin and epirubicin at 30 mg/mq, gemcitabine at 800 mg/mq and capecitabine at 1250 mg/mq/day per os for 14 days every 14 days for 6 months
  Interventions: Drug: capecitabine; Drug: cisplatin; Drug: epirubicin; Drug: gemcitabine
- perioperative PEXG (Experimental): cisplatin and epirubicin at 30 mg/mq, gemcitabine at 800 mg/mq and capecitabine at 1250 mg/mq/day per os for 14 days every 14 days for 3 months before surgery and 3 months after surgery
  Interventions: Drug: capecitabine; Drug: cisplatin; Drug: epirubicin; Drug: gemcitabine
- Adjuvant Gemcitabine (Active Comparator): Adjuvant Gemcitabine at 1000 mg/mq for 3 weeks every 4 weeks for 6 months
  Interventions: Drug: gemcitabine

INTERVENTIONS:
Drug: capecitabine — 1250 mg/mq/day per os for 14 days every 14 days for 6 months
  Other Names: XELODA
  Arms: adjuvant PEXG; perioperative PEXG
Drug: cisplatin — 30 mg/mq every 14 days for 6 months
  Other Names: cisplatino TEVA
  Arms: adjuvant PEXG; perioperative PEXG
Drug: epirubicin — 30 mg/mq every 14 days for 6 months
  Other Names: farmorubicina
  Arms: adjuvant PEXG; perioperative PEXG
Drug: gemcitabine — ARM A: 1000 mg/mq for 3 weekly infusions every 4 weeks for 6 months ARM B and C: 800 mg/mq every 14 days for 6 months
  Other Names: GEMZAR

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as gemcitabine hydrochloride, cisplatin, epirubicin hydrochloride, and capecitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving gemcitabine hydrochloride, with or without cisplatin, epirubicin hydrochloride, and capecitabine before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed. Giving these drugs after surgery may kill any tumor cells that remain after surgery.

PURPOSE: This randomized phase II/III trial is studying how well gemcitabine hydrochloride, with or without cisplatin, epirubicin hydrochloride, and capecitabine, works when given before and/or after surgery in treating patients with stage I or stage II pancreatic cancer that can be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess the proportion of patients who are event-free (defined as disease progression, local recurrence, distant metastasis, new tumor, or death) at 1 year after neoadjuvant therapy comprising gemcitabine hydrochloride with cisplatin, epirubicin hydrochloride, and capecitabine (PEXG), and adjuvant chemotherapy comprising gemcitabine hydrochloride or PEXG regimen in patients with resectable stage I or II adenocarcinoma of the pancreas. (phase II)
* To assess whether the best experimental regimen, which will be selected on the basis of the phase II part of the trial, is able to improve overall survival when compared to standard adjuvant gemcitabine in these patients. (phase III)

Secondary

* To assess radiological, biochemical, and pathological response rate (neoadjuvant arm only) in these patients.
* To assess surgical resection rate, surgical mortality and morbidity, and proportion of patients with negative surgical margins.
* To assess lymph node status in these patients.
* To determine tolerability of these regimens in these patients.

OUTLINE: This is a multicenter study. Patients are stratified according to center. Patients are randomized to 1 of 3 treatment arms.

* Arm I (adjuvant gemcitabine hydrochloride) : Patients receive gemcitabine hydrochloride IV over 1 hour on days 1, 8, and 15. Courses repeat every 28 days for 6 months in the absence of disease progression or unacceptable toxicity.
* Arm II (adjuvant cisplatin, epirubicin hydrochloride, gemcitabine hydrochloride, and capecitabine [PEXG regimen]): Patients receive cisplatin IV over 1 hour on days 1-5, epirubicin hydrochloride IV on days 1 and 8, gemcitabine hydrochloride IV over 1 hour on days 1 and 8, and oral capecitabine on days 1-14. Treatment repeats every 14 days for 6 months in the absence of disease progression or unacceptable toxicity.
* Arm III (neoadjuvant and adjuvant PEXG regimen): Patients receive neoadjuvant cisplatin IV over 1 hour on days 1-5, epirubicin hydrochloride IV on days 1 and 8, gemcitabine hydrochloride IV over 1 hour on days 1 and 8, and oral capecitabine on days 1-14. Treatment repeats every 14 days for up to 3 months. Patients then undergo surgery for pancreatic cancer followed by adjuvant (within 2 months of surgery) PEXG given as in neoadjuvant therapy. Treatment with adjuvant PEXG repeats every 14 days for 3 months in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 1 year, every 4 months for 2 years, and then every 6 months thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically* confirmed adenocarcinoma of pancreas

  * Stage I-II disease
  * Resectable disease
* No superior mesenteric vein or artery, portal vein, celiac trunk, or hepatic artery infiltration
* No symptomatic duodenal stenosis
* NOTE: Patients without histological or cytological results may be allowed provided ≥ 1 attempt has been made by needle aspiration with negative imaging and clinical signs suggestive of adenocarcinoma.

PATIENT CHARACTERISTICS:

* Karnofsky performance status 70-100%
* WBC ≥ 3,500/mm³
* ANC ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 10 g/dL
* Creatinine ≤ 1.5 mg/dL
* ALT and AST ≤ 3 times upper limit of normal
* Bilirubin ≤ 3 mg/dL
* No prior or concurrent malignancy within the past 5 years except for surgically cured carcinoma in situ of the cervix or basal cell or squamous cell carcinoma of the skin
* Not pregnant or nursing
* No psychological, familial, sociological, or geographical condition that would potentially hinder study compliance or follow-up schedule

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy or radiotherapy for pancreatic adenocarcinoma
* No other concurrent experimental drugs

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2010-05; Primary Completion 2017-04 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Event-free survival at 1 year (phase II) | every 3 months
  CT scan

SECONDARY OUTCOMES:
Radiological, biochemical, and pathological response rate (neoadjuvant arm only) | after 3 months of induction therapy
  CT scan, CA19.9 serology; pathology report
Surgical resection rate | immediately after surgery
  surgeon report
Surgical mortality and morbidity | immediately after surgery
  surgeon report
Tolerability | every 2 weeks during therapy
  outpatient visit; laboratory report
Proportion of patients with negative surgical margins | immediately after surgery
  pathology report
Lymph node status | immediately after surgery
  pathology report

CONTACTS AND LOCATIONS:
Overall Officials: Michele Reni, MD, Principal Investigator — Istituto Scientifico H. San Raffaele
Locations (1):
- Istituto Scientifico H. San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Reni M, Balzano G, Zanon S, Zerbi A, Rimassa L, Castoldi R, Pinelli D, Mosconi S, Doglioni C, Chiaravalli M, Pircher C, Arcidiacono PG, Torri V, Maggiora P, Ceraulo D, Falconi M, Gianni L. Safety and efficacy of preoperative or postoperative chemotherapy for resectable pancreatic adenocarcinoma (PACT-15): a randomised, open-label, phase 2-3 trial. Lancet Gastroenterol Hepatol. 2018 Jun;3(6):413-423. doi: 10.1016/S2468-1253(18)30081-5. Epub 2018 Apr 4. PMID 29625841